CLINICAL TRIAL: NCT00588081
Title: Immediate Vaginal Reconstruction Following Oncologic Resection: Surgical Outcomes, Patient Satisfaction and Sexual Function
Brief Title: Immediate Vaginal Reconstruction After Oncologic Resection: Surgical Outcomes, Patient Satisfaction and Sexual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-044
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Vaginal Cancer
Keywords: Vaginal Reconstruction
MeSH Terms: conditions — Vaginal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Participants will receive a cover letter, questionnaire and invitation to participate in a post-operative interview.
  Interventions: Behavioral: QOL

INTERVENTIONS:
Behavioral: QOL — Those women who chose to have an interview will be scheduled for a 45 to 60 minute open-ended interview with a trained research assistant and sign consent at the time of the interview.

SUMMARY:
This study is being done to find out more about the experience women have with vaginal reconstruction. We hope to learn about their quality of life, sexual function, and body image. We would like to find out how happy women are with surgery. We also want to know what things should be changed or improved. Since you have had this surgery, we would like to ask you to take part in an interview.

DETAILED DESCRIPTION:
The purpose of this study, entitled immediate vaginal reconstruction following oncologic resection: Surgical outcomes, patient satisfaction and sexual function is to determine postoperative complications, patient satisfaction, quality of life and level of sexual functioning among patients who have undergone vaginal reconstruction following tumor resection and/or pelvic exenteration.This study will have three components: 1) a chart review to determine postoperative complications and anatomic characteristics of the neo-vagina, 2) a postoperative questionnaire consisting of validated survey instruments to assess quality of life, body image and sexual function and 3) a postoperative qualitative interview to examine quality of life after vaginal reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Immediate partial or total vaginal reconstruction with myocutaneous or fasciocutaneous flaps, following pelvic exenteration or tumor resection at MSKCC during the study period from January 1, 1993 to, March 30, 2007.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To determine perioperative and postoperative complication rates among patients having undergone immediate vaginal reconstruction following tumor resection and/or pelvic exenteration. | A single questionnaire and or interview

SECONDARY OUTCOMES:
To determine patient satisfaction, quality of life and level of sexual functioning among patients having undergone immediate vaginal reconstruction following tumor resection and/or pelvic exenteration. | Single Questionnaire and or interview
To determine the physical adequacy of the neo-vagina among patients having undergone immediate vaginal reconstruction following tumor resection and/or pelvic exenteration. | A single questionnaire and or interview

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pusic, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center website — http://www.mskcc.org